CLINICAL TRIAL: NCT03177057
Title: Self-Monitoring and Readiness Texting Project (SMART)
Brief Title: SMART Project in Preventing Skin Cancer
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Carolyn Heckman, Principal Investigator, Fox Chase Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB12846; NCI-2015-02089 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB12846 (Other: Fox Chase Cancer Center); P30CA006927 (NIH)
Record Dates: First submitted 2017-06-02; First posted 2017-06-06 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Skin Carcinoma

ARMS (4):
- Arm I (self-monitoring) (Experimental): ARM I (SELF-MONITORING): Patients complete tanning and sun protection usage entries daily for 14 days.
  Interventions: Behavioral: Compliance Monitoring; Other: Questionnaire Administration
- Arm II (text messages) (Experimental): ARM II (TEXT MESSAGES): Patients receive individualized text messages based on baseline assessment of tanning motives (appearance, enjoyment, social) daily for 14 days.
  Interventions: Other: Health Telemonitoring; Other: Questionnaire Administration
- Arm III (self-monitoring, text messages) (Experimental): ARM III (COMBINED GROUP): Patients complete tanning and sun protection usage entries and also receive individualized text messages daily for 14 days.
  Interventions: Behavioral: Compliance Monitoring; Other: Health Telemonitoring; Other: Questionnaire Administration
- Arm IV (questionnaire administration) (Sham Comparator): ARM IV (CONTROL GROUP): Patients complete study assessments.
  Interventions: Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Compliance Monitoring — Record behavior
  Arms: Arm I (self-monitoring); Arm III (self-monitoring, text messages)
Other: Health Telemonitoring — Receive health monitoring text messages
  Arms: Arm II (text messages); Arm III (self-monitoring, text messages)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This pilot clinical trial studies how well Self Monitoring And Readiness Texting (SMART) project works in sun exposure and protection behaviors. Measuring how behavior tracking and individually tailored messages affect risk behaviors in patients with skin cancer may help doctors plan the best prevention plan and decrease national melanoma incidence and mortality.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test the effects of a behavior tracking and individually-tailored daily text message intervention on sun protection and exposure behaviors and to see if these techniques will be most effective in conjunction or separately.

SECONDARY OBJECTIVES:

I. To examine mediators in the effects of the intervention on safe sun behaviors, based on Fishbein?s Integrative Model.

OUTLINE: Patients are randomized to 1 of 4 study arms.

ARM I (SELF-MONITORING): Patients complete tanning and sun protection usage entries daily for 14 days.

ARM II (TEXT MESSAGES): Patients receive individualized text messages based on baseline assessment of tanning motives (appearance, enjoyment, social) daily for 14 days.

ARM III (COMBINED GROUP): Patients complete tanning and sun protection usage entries and also receive individualized text messages daily for 14 days.

ARM IV (CONTROL GROUP): Patients complete study assessments.

After completion of study, patients are followed up at 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Women from the Philadelphia metropolitan area who own a mobile phone and who meet criteria for at least moderate risk of skin cancer based on a brief risk assessment tool

Ages: 18 Years to 29 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2013-04-23 (Actual); Primary Completion 2014-07-30 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Change in ultraviolet radiation (UV) exposure and sun protection behaviors based on behavior tracking and individually tailored daily text messages | Baseline to up to 2 weeks
  Multiple variable regression models will be performed to examine the effect of the intervention on the outcomes. All post-baseline outcomes will be used as dependent variables. The baseline scores, intervention group, and time of the assessment will be included. To account for the within subject correlation of the responses, we will fit the model using Generalized Estimating Equations assuming an autoregressive working correlation matrix for each subject. Any p-value from the pairwise comparison that is less than 0.05 will be considered worthy of further study.

SECONDARY OUTCOMES:
Mediators and moderators of the intervention on behavior | At 2 weeks
  Mediation will be assessed by examining indirect effects, with bootstrapped confidence intervals to be calculated around the mediated effects. For participants who use the self-monitoring app, hierarchical linear modeling will be used to examine associations between tanning and sun protection as they occur daily, and motives for doing so. Using lagged multi-level models, the within-person model allows for assessment of individual change in behavior over the two-week time period, as well as the effect of each day?s behavior on behavior occurring on subsequent days. The between-person model allo

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Heckman, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States